CLINICAL TRIAL: NCT04755322
Title: Hydroxychloroquine is an Immunomodulator for Improvement of Pregnancy Outcomes in Preeclampsia
Brief Title: Hydroxychloroquine in Prevention of Preeclampsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mahmoud Mohammed, Assisstant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HPP_2020
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Hydroxychloroquine; Folic Acid; Aspirin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hydroxychloroquine group (Other): hydroxychloroquine 400 mg+ Folic Acid 5 mg+ Low-dose aspirin 75 mg
  Interventions: Drug: Hydroxychloroquine; Drug: Folic acid; Drug: Low-dose aspirin
- control group (Other): Folic Acid 5 mg+ Low-dose aspirin 75 mg
  Interventions: Drug: Folic acid; Drug: Low-dose aspirin

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine 400 mg at start of pregnancy
  Arms: hydroxychloroquine group
Drug: Folic acid — 5 mg
Drug: Low-dose aspirin — 75 mg

SUMMARY:
Pre-eclampsia complicates up to 8% of pregnancies and is a major contributor to maternal mortality and morbidity The only effective treatment is delivery, which leads to significant neonatal morbidity and mortality if carried out preterm, especially when the disease occurs early in pregnancy. Vascular endothelial dysfunction and immunological impairment are associated with preeclampsia. To date, there is no effective or optimal therapeutic approach for these conditions. Hydroxychloroquine has endothelial protective action via ant diabetic, lipid lowering, antioxidant effects or direct endothelial protection. Hydroxychloroquine is an antimalarial and immunomodulatory agent. In pregnancy, hydroxychloroquine is prescribed for inflammatory conditions associated with adverse perinatal outcomes such as systemic lupus erythematosus, antiphospholipid syndrome and placental inflammatory lesions such as chronic histiocytic intervillositis, hydroxychloroquine has therapeutic potential to improve placental function in pregnancies associated with heightened inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women in 1st 6 weeks gestation.
2. History of preeclampsia in previous pregnancies.
3. Women who accepted to participate

Exclusion Criteria:

1. Risk factors (multiple gestation, chronic hypertension, chronic renal disease).
2. Known contraindication to a treatment by HCQ (retinopathy, hypersensitivity to chloroquine or HCQ, G6PD deficiency, chronic liver or kidney insufficiency, heart block, significant chronic digestive, hematologic disease epilepsy or psychotic disorders.) or disorder of lactose metabolism
3. Patient already using HCQ (rheumatoid arthritis, Lupus, solar eczema). 4.impossible for follow up

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
number of cases of preeclampsia | 9 month

SECONDARY OUTCOMES:
number of cases of Number of pregnancy complications such as FGR, IUFD, and gestational hypertension, HELLP syndrome, placental abruption, eclampsia, ICU admission and pulmonary edema | 9 month
Number of pregnancies with fetal malformation | 9 months
number of live birth | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Abdel-rahman Mahmoud Mohammed, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided